CLINICAL TRIAL: NCT02251106
Title: Effect of Lumbar Bracing on Spinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Aspen Medical Products (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00030976
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- -LBP/-Brace (No Intervention): Subjects in this arm did not have back pain nor did they wear brace (asymptomatic controls). Subjects had their spine function measured before and after a two week period.
- -LBP/+Brace (Active Comparator): Intervention = Lumbar corset (Quickdraw, Aspen Medical Products) Subjects in this arm did not have back pain but wore a brace for a two week period (asymptomatic intervention). Subjects had their spine function measured before and after a two week period.
  Interventions: Device: Lumbar corset (Quickdraw, Aspen Medical Products)
- +LBP/+Brace (Experimental): Intervention = Lumbar corset (Quickdraw, Aspen Medical Products) Subjects in this arm had back pain and wore a brace for a two week period (symptomatic intervention). Subjects had their spine function measured before and after a two week period.
  Interventions: Device: Lumbar corset (Quickdraw, Aspen Medical Products)

INTERVENTIONS:
Device: Lumbar corset (Quickdraw, Aspen Medical Products) — The corset (a.k.a. brace) is made of webbing and elastic. It is wrapped around the trunk and tightened with Velcro and a series of cords (like tying shoes).
  Other Names: Soft lumbar brace
  Arms: +LBP/+Brace; -LBP/+Brace

SUMMARY:
A recent province-wide survey (Alberta, Canada) suggests that clinicians' beliefs about soft lumbar bracing for low back pain (LBP) vary substantially. Approximately 50% of clinicians (MDs, DCs, PTs) find back braces "useful" for acute back pain while the remaining half report that bracing causes muscle atrophy. While previous studies suggest bracing for acute low back conditions can reduce pain and does not cause atrophy, no prior study has assessed back function after bracing using self-reported and objective measures within the same cohort.

PURPOSE:

To assess both self-reported and objective measures of spine function before, and after, use of an inelastic lumbar brace over a two week period.

STUDY DESIGN:

Before-After Design

OUTCOME MEASURES:

Self-reported spine function, spinal stiffness and muscle endurance.

METHODS:

Three groups were studied: asymptomatics who did not wear a brace (-LBP/-Brace), asymptomatics who were braced (-LBP/+Brace) and acute LBP subjects who were braced (+LBP/+Brace). Both groups of braced subjects (-LBP/+Brace; +LBP/+Brace) were instructed to wear the brace continually for 2 weeks with the exception of bedroom & bathroom activities. Before and after the 2 week period, 3 measures of spine function were performed: spinal stiffness via motorized indentation of the L3 spinous process, a modified Sorensen test (timed lumbar extension against gravity), and the Oswestry Disability Index (ODI). Unbraced (-LBP/-Brace) subjects were studied over the same time with the same measures. Repeated measures analyses of variance were conducted for all three outcomes with a significance level of 0.05.

DETAILED DESCRIPTION:
Background: While various treatments for low back pain (LBP) are prescribed, one in particular appears to be frequently self-prescribed: external lumbar bracing (i.e. elastic corsets and other similar devices). Given that the mechanical function of the back is to bear static and dynamic loads and that most LBP is thought to be mechanical in nature, there is a biological plausibility that underlies bracing as a treatment for LBP Indeed, several reports suggest lumbar bracing may be effective for some LBP patients.

The high frequency of self-prescribed bracing may be the result of the clinical community's reluctance to prescribe these devices. Approximately half of Alberta spine clinicians believe that spine bracing results in muscle atrophy and/or future dependency on braces. Conversely, recent work from our laboratory has shown that after two weeks of brace wearing, the volume of spinal muscles remains unchanged in asymptomatic subjects (i.e. no brace-induced atrophy was caused)

Objective and hypothesis: While bracing for 14 days does not result in decreased muscle volume in asymptomatic subjects, there is a need to understand if bracing preserves muscle volume while muscle function declines. This information would allow us to understand the effects of bracing on spinal function independent of changes in muscle volume. Therefore, we hypothesize that that brace-wearing will result in an insignificant alteration in spinal function.

Future Relevance: Results from this pilot study will allow us to construct future investigations to reveal the underlying mechanisms of bracing with respect to the alleviation of LBP.

Subjects: Subjects of both genders between the ages of 18 and 65 will be recruited from the University of Alberta and surrounding area. The target recruitment populations are 1) asymptomatic subjects and 2) those with low back pain. Subjects excluded from the study will have a history of back pain with red flags, those who are pregnant (or believe they may be pregnant) or other contraindications described in the full protocol.

Methods: Potential subjects will complete a survey to obtain demographic data as well as a focused medical history and physical examination performed by one of the research team. If a subject meets the inclusion/exclusion criteria and provides written, informed consent, they will be enrolled in the study. Those not able to be enrolled will be thanked and dismissed.

Asymptomatic subjects will be assigned randomly into a brace and non-brace cohort. From the recruited subjects, three cohorts will be created: 1) Asymptomatic subjects who will wear a brace (-LBP/Brace+), 2) asymptomatic subjects who will not wear a brace (-LBP/-Brace) and 3) low back pain subjects who will wear a brace (+LBP/+Brace). Because this experiment is not designed to assess brace efficacy, there is no need to include a cohort of symptomatic subjects who do not wear a brace. Each subject who will wear a brace will be fitted and sized for an elastic brace supplied at no charge to the subject. Subjects will be instructed on how to don and remove the brace as well as the circumstances when they are permitted to remove the brace (washroom, shower, sleep). The subject will also be informed that the brace has a monitoring feature to determine brace compliance as well as their activity level.

As soon as possible after brace fitting, a battery of tests will be conducted to determine each subject's spinal function. These tests are as follows:

1. The Oswestry Disability Index (OWDI). The OWDI is a self-reported measure of function. The OWDI has established reliability and validity and has been used extensively in low back pain research.
2. Spinal Stiffness testing. This test uses a blunt probe to push into the back of a resting subject to measure the stiffness of the spine. It was developed in our lab and has been used in many prior studies both at the Universities of Alberta, Hong Kong and Utah.
3. Rehabilitation Ultrasound Imaging (RUSI). This test uses ultrasound to image spine muscles during simple tasks (e.g. arm raising) to quantify the ability of the back muscles to contract with the desired magnitude and timing. This test is well-described in the literature and has been approved for use previously in our laboratory.
4. Modified Sorensen test. This is a timed test of spine function where subjects are asked to straighten their backs from a semi-inclined position until pain onset and/or failure to maintain the target position. The test, and its variants, has been well-studied since it was first described in 1984. The modified version of the test to be used here has been shown to be safe to perform in acute back pain subjects.

The subject will now be released to their usual activities of daily living for a period of 14 days.

To determine if there are any problems in subjects wearing braces, those subjects will be contacted by the PI or research team within the first 24 hours following brace fitting and then approximately every three days after that time. If a correction to the brace cannot be made that is satisfactory to the research team and the subject, the subject will thanked and dismissed.

Following the two week experiment period, subjects will attend the laboratory. Usage data will then be extracted from the data logger of those wearing braces. If the subject has worn the brace for less than 75% of the requested time, the subject will be dismissed and thanked for their participation. If subjects have worn the brace for more than 75% of the requested time, the spinal function tests will be performed for a second time.

Change scores of each of the 5 spine function tests will be calculated and then compared between the three cohort using an analysis of variance (alpha = 0.05).

Expected results: Given our prior data that muscle volume does not changes after 14 days of bed rest, it is expected that brace-wearing will not reduce spinal function in symptomatic or asymptomatic populations.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the study will be between the ages of 18 and 65 and include both genders.

Asymptomatic subjects will be asymptomatic for low back pain for a period of 3 months or more.

Symptomatic subjects will have non-specific low back pain that is of an acute or chronic nature. Recruiting those with non-specific low back pain ensures that we are not enrolling subjects with a specific cause for back pain (eg, spinal fracture) for which spinal function testing is contraindicated.

Exclusion Criteria:

Specific to the spinal function tests used here, excluded subjects will include those with suspected or confirmed malignancy as the cause for back pain, spinal fracture (current or within the last 5 years), previous non-day surgery to the abdomen, spine pelvis or hips, presence of nerve root involvement (presence of at least 2 of the 3: myotomal weakness, altered sensation in dermatomal patterns, and/or altered knee/ankle reflexes), ankylosing spondylitis and current skin conditions that may be aggravated by bracing, These exclusion criteria relate to back conditions for which spinal function testing is contraindicated (eg, malignancy) or in which there is a greater chance of causing discomfort (eg, nerve root involvement).

General exclusion criteria include: osteoporosis, rheumatoid arthritis (or taking any disease modifying anti-rheumatic drugs), pregnancy or suspected pregnancy, known severe spondylolisthesis, severe scoliosis, Type I diabetes mellitus, hyperparathyroidism, hyperthyroidism, inability to lie prone for at least 40 minutes, inability to tolerate back extension or spinal indentation (eg, indentations cause discomfort), inability to speak or read English (to ensure that participants understand what is happening and can reliably relay any discomfort). People currently taking muscle relaxants will also be excluded. In addition, subjects who are hypertensive, or are prone to hypertension (smokers), will be excluded from this study as will subjects who have a history of aortic aneurysm. Although hypertension and aortic aneurysm are not contraindications to lumbar bracing, we will exclude them from this trial. Finally, some persons with low or high body mass indexes may not be eligible to participate if they are unable to be fitted properly with a brace. Subjects will also be excluded if they feel they would be unable to lie prone (i.e. face-down) for up to 1 hour during spinal stiffness and RUSI testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg N Kawchuk, PhD, Principal Investigator — University of Alberta

RESULTS

PARTICIPANT FLOW:
Groups:
- -LBP/-Brace: No brace. Subjects in this arm did not have back pain nor did they wear a brace (asymptomatic controls).
- -LBP/+Brace: Intervention = Lumbar corset (Quickdraw, Aspen Medical Products) Subjects in this arm did not have back pain but wore a brace for a two-week period (asymptomatic intervention). Subjects had their spine function measured before and after a two-week period.
- +LBP/+Brace: Intervention = Lumbar corset (Quickdraw, Aspen Medical Products) Subjects in this arm had back pain and wore a brace for a two-week period (symptomatic intervention). Subjects had their spine function measured before and after a two-week period.
Period: Overall Study
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace
Started | 19 | 18 | 17
Completed | 19 | 18 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace | Total
Number analyzed (Participants) | 19 | 18 | 17 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 17 | 54
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (15.3) | 33.1 (12.9) | 39.2 (12.0) | 36.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 9 | 26
  Male | 11 | 9 | 8 | 28
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 18 | 17 | 54
Oswestry Disability Index [Mean (Standard Deviation); unit: units on a scale] — The Oswestry Disability Index (ODI) questionnaire is a self-reported measure of function that examines perceived level of disability in 10 everyday activities of daily living.
  The 6 statements are scored from 0 to 5 (mild to worst imaginable.
  If all 10 sections are completed the ODI score is calculated as follows:
  (Total scored) out of 50 (total possible score) x 100 = __%
  If one section is missed (or not applicable) the score is calculated:
  (Total scored) / (total possible score with section removed) x 100 = __%
  units on a scale | .42 (.9) | .83 (1.76) | 10.41 (5.87) | 3.08 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) questionnaire is a self-reported measure of function that examines the perceived level of disability.
  The ODI is made up of 10 questions. Each question is scored from 0-5 (minimum to maximum)
  The point total from each section is summed and then divided by the total number of questions answered and multiplied by 100 to create a percentage disability. The scores range from 0-100% with lower scores meaning less disability.
  If one section is missed (or not applicable) the score is calculated:
  (Total scored) / (total possible score with section removed) x 100 = __%
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace | -LBP/-Brace @ 2 Weeks | -LBP/+Brace @ 2 Weeks | +LBP/+Brace @ 2 Weeks
Number analyzed (Participants) | 19 | 18 | 17 | 19 | 18 | 17
score on a scale | .42 (.9) | .83 (1.76) | 10.41 (5.87) | .42 (1.02) | .52 (1.31) | 6.1 (5.62)

2. Secondary Outcome: Modified Sorensen Test
Description: This is a timed test of spine endurance where subjects are asked to straighten their backs from a semi-prone position. In patients who experience no difficulty in holding the position, the test is stopped after 240s. A position-holding time less than 176 seconds predicts low back pain during the next year in males, whereas a time greater than 198 seconds predicts absence of low back pain.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- -LBP/+Brace: Intervention = Lumbar corset (Quickdraw, Aspen Medical Products) Subjects in this arm did not have back pain but wore a brace for a two week period (asymptomatic intervention). Subjects had their spine function measured before and after a two week period.
  .
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace | -LBP/-Brace @ 2 Weeks | -LBP/+Brace @ 2 Weeks | +LBP/+Brace @ 2 Weeks
Number analyzed (Participants) | 19 | 18 | 17 | 19 | 18 | 17
seconds | 96.47 (62.61) | 119.83 (84.07) | 49.76 (23.67) | 119.21 (65.48) | 129.00 (88.14) | 54.35 (30.59)

3. Secondary Outcome: Bulk Spinal Stiffness
Description: This test uses a blunt probe to non-invasively push into the back of a prone, resting subject.
Time Frame: 2 weeks
Population: Outcome measure not assessed.
Groups:
- -LBP/-Brace: No brace Subjects in this arm did not have back pain nor did they wear a brace (asymptomatic controls).
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Rehabilitation Ultrasound Imaging
Description: This test uses ultrasonic imaging to visualize spine muscles during simple tasks such as arm extension
Time Frame: 2 weeks
Population: Outcome measure not assessed.
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were defined as any adverse experience occurring during the course of the study.
  Adverse events could be reported at any time by the participants who were additionally asked directly about adverse events in their last face to face session.
Arm/Group | -LBP/-Brace | -LBP/+Brace | +LBP/+Brace
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No